CLINICAL TRIAL: NCT04319354
Title: Evaluation of cfDNA as a Marker of Response to Neoadjuvant Chemoradiotherapy in Locally Advanced Rectal Cancer
Brief Title: Evaluation of cfDNA as a Marker of Response in Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Pedro Hispano (Other)
Collaborators: Diogo Melo Pinto, MD, Hospital Pedro Hispano (Unknown); Telma Fonseca, MD, Centro Hospitalar de São João (Unknown); Silvestre Carneiro, PhD, Centro Hospitalar de São João (Unknown); Isabel Prieto, PhD, Hospital La Paz, Madrid (Unknown)
Responsible Party: Principal Investigator, Marina Morais, Principal Investigator, Hospital Pedro Hispano
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 85/19/56C
Record Dates: First submitted 2020-03-09; First posted 2020-03-24 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Cancer of Rectum
Keywords: rectal cancer; neoadjuvant therapy; cfDNA
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pCR (Experimental)
  Interventions: Diagnostic Test: Analysis of cfDNA
- Partial responders (Experimental)
  Interventions: Diagnostic Test: Analysis of cfDNA
- Non-responders (Active Comparator)
  Interventions: Diagnostic Test: Analysis of cfDNA

INTERVENTIONS:
Diagnostic Test: Analysis of cfDNA — Analysis of cfDNA through liquid biopsy

SUMMARY:
A pathological complete response (pCR) after surgery occurs in approximately 20% of rectal cancer patients submitted to neoadjuvant chemotherapy, with apparent survival benefit. This group could, potentially, be spared the morbidity of surgery.

The diversified response to neoadjuvant chemotherapy (nCRT) amongst tumors suggests a complex relationship between tumor biology and response possibly due to a number of genetic or molecular pathways that might regulate chemoradiosensitivity.

Accumulating evidence indicated that circulating cell-free nucleic acids can be a promising biomarker of response, in liquid biopsy, for rectal cancer. The concentration of baseline plasma cell-free DNA (cfDNA) appears significantly higher in responders compared to non-responders.

The objective of this study is to investigate the potential role of cfDNA as a marker of pCR (or partial response) to nCRT as well as a marker of outcomes (overall survival and disease-free survival).

The investigators are conducting a prospective, observational, cohort, non-randomized study of consecutive patients with locally advanced rectal cancer submitted to nCRT, followed by surgical excision 6-12 weeks later. Patients are assigned to groups according to their pathological response to nCRT. A total of 20 patients with complete pathological response, 50 partial response and 50 non-responders will be selected over a year and followed for another year. Participants will be observed and examined during the entire course of treatment and the follow-up period.

Serial analysis of cfDNA through liquid biopsies will be performed in consecutive patients at specific time points (pre-nCRT, post-nCRT and postoperative week 1), incorporating analysis of concentration, dimension of DNA fragments, % of mutation frequency (CIN, APC, p53, MSI, KRAS, BRAF, EGFR, cKIT) and next-generation sequencing of tumour biopsy and surgical specimens.

This study will serve as the feasibility of a larger, comparative study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18 years old, ECOG 0-2
2. High-risk patients with biopsy proven rectal adenocarcinoma who will undergo long-course chemoradiotherapy and who are potentially eligible for curative surgery
3. Patients who can fully understand the content of the informed consent form and sign it upon their own opinion
4. Patients who can coordinate with the researchers to undergo the long-term post-treatment rechecks and follow-up

Exclusion Criteria:

1. Patient has any underlying or current medical condition, which would interfere with the evaluation of the patient (e.g., end-stage liver disease, pulmonary hypertension, systemic lupus erythematosus etc.).
2. Patient has severe mental illness.
3. Patient has any other conditions, which would interfere with the evaluation of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Ryan tumor regression grade system (number of patients with complete/partial/no response) | Through study completion, an average of 1 year
  Tumour pathological response, on surgical specimen, to neoadjuvant chemoradiotherapy

SECONDARY OUTCOMES:
Number of participants with 1 and 2-year disease free recurrence | 1 and 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pedro Hispano, Matosinhos Municipality, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: since the beginning, for 2 years